CLINICAL TRIAL: NCT00290160
Title: The Effect of Early Protein Supplementation on Prevention of Hyperkalemia in Extremely Low Birth Weight Infants
Brief Title: Early Protein Supplementation on Prevention of Hyperkalemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 012-9000-400
Record Dates: First submitted 2006-02-08; First posted 2006-02-10 (Estimated); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Hyperkalemia
Keywords: Hyperkalemia; Protein; Hyperglycemia; ELBW
MeSH Terms: conditions — Hyperkalemia; Hyperglycemia

INTERVENTIONS:
Behavioral: Protein supplementation

SUMMARY:
Evaluate if early protein supplementation decreases the incidence of hyperkalemia in Extremely Low Birth Weight Infants (babies less than 1,000 grams birth weight).

DETAILED DESCRIPTION:
Randomized double blind prospective clinical trial. All infants admitted to University Hospital neonatal intensive care unit with birth weight of < 1000 grams, mmore than 24 weeks gestation and with no congenital anomalies will be enrolled in the study. This will include inborn infants and those that are transported from outlying hospitals and admitted at <12 hours of life. After informed consent, infants will be randomized to receive either standard of care nutritional management or nutritional management per study protocol with the addition of protein supplementation. Randomization will take place in the pharmacy.

Control Group: Infants enrolled in the control group will be started on intravenous fluids (IVF) on admission to the NICU with 5% Dextrose and 1500 mg calcium gluconate per 500 cc for a total fluid intake of either 120 or 150 cc/kg/day. The attending neonatologist in accordance with the infant's gestational age and maturity will make the decision regarding total fluid intake. The control group will be started at 0.5 gram/kg/d of protein ( Amynosin PF) on DOL 1 and increase by 0.5 gram/kg/day every day to a maximum of 3 grams/kg/day.

Study group: The study group will receive the same total fluid intake (120 cc/kg/day or 150 cc/kg/day) and 5% dextrose infusion with calcium gluconate and the addition of 2 grams/kg/day of protein (Aminosyn PF). The study group will receive 2 grams/kg/day of protein for 24 hours to 36 hours and will increase by 1 gram/kg/day up to a maximum of 4 grams/kg/day.

In both groups, caloric intake will start at 29-34 kcal/kg day (i.e., approximately 20-25 calories per kilogram from glucose and 9 calories per kilogram from lipids). Caloric intake will be progressively increased depending on the infant's tolerance to glucose. Protein to glucose ratio in the control group will be 250-312 and nitrogen balance ratio (including all calories) will be approximately 362-425. In the study group, protein to glucose ratio will be 64-80 and nitrogen balance ratio (including all calories) will be 93-109. The control group corresponds to the current standard of care. The study group nitrogen balance is within the limits of recent studies which show that a nitrogen balance ratio of 46-78 is appropriate for ELBW infants.

Glucose infusion rate (GIR) will be increased by attending neonatologist depending on infant's glucose tolerance. Usually GIR is started at 6 mg/kg/min and increased by 1 milligram per kilo per minute every 24 hrs. in ELBW infants. For fluctuations in glucose, adjustments in glucose infusion rate (GIR) will be via piggyback dextrose to the IVF if necessary.

Lipids will be supplied as a 20% solution and will be started by attending neonatologist according to standard of care (0.5-1 gr/kg first day of life, then increases of 0.5-1 gr/kg per day up to a maximum of 3 gr/kg day).

All infants will be started on Total Parenteral Nutrition (TPN) on DOL 1. The amino acid solution (Aminosyn PF) will be supplemented with 40 mg cysteine hydrochloride/kg/day in both groups since it is considered to be one of the essential amino acids for premature infants. Stable isotope studies have suggested improved protein retention with cysteine supplementation. 3 The amino acid solution will be added via pharmacy per study protocol. Subjects will continue to receive supplementation for the first week of life.

Initiation of feedings, TPN, fluid, and electrolyte intake will be determined by the attending neonatologist.

If the infant develops hyperkalemia (>6.5 mmol/lt), treatment will be determined by attending neonatologist based on standard of care incluiding: an increase in intravenous fluid delivery, diuretic therapy (lasix), correction of acidosis, close monitoring of ionized and total calcium levels and correction with calcium gluconate if needed, glucose and insulin infusion , kayexalate, and if refractory, exchange transfusion might be considered.

Following completion of the study, we will continue to monitor standard laboratory data, including serum and urine electrolytes. We will also monitor growth until hospital discharge. Following discharge, infants will be followed in PREMIEre clinic for neurodevelopmental outcome with Bayley testing at 6, 12, and 18 months CGA. In addition to the primary outcome reduction in incidence of hyperkalemia, our secondary outcomes of interest include the incidence of hyperglycemia, the incidence of periventricular-intraventricular hemorrhage (PIVH), renal function, growth, and neurodevelopmental outcome at 18 months corrected gestational age.

ELIGIBILITY:
Inclusion Criteria: ELBW infants with birth weight <1000 grams . Enrollment within the first 12 hr of life.

Exclusion Criteria: major congenital anomalies; gestational age less than 24 weeks, infants not resuscitated, death.

Ages: 1 Minute to 12 Hours | Sex: All
Age Groups: Child
Enrollment: 62
Dates: Start 2002-12; Primary Completion 2005-09 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Incidence of hyperkalemia in between groups

SECONDARY OUTCOMES:
Incidence of hyperglycemia, post-natal growth, neurodevelopmental outcome at 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia L Blanco, MD, Principal Investigator — University of Texas
Locations (1):
- University Health System, San Antonio, Texas, United States

REFERENCES:
- [Derived] Blanco CL, Gong AK, Schoolfield J, Green BK, Daniels W, Liechty EA, Ramamurthy R. Impact of early and high amino acid supplementation on ELBW infants at 2 years. J Pediatr Gastroenterol Nutr. 2012 May;54(5):601-7. doi: 10.1097/MPG.0b013e31824887a0. PMID 22228000
- [Derived] Blanco CL, Gong AK, Green BK, Falck A, Schoolfield J, Liechty EA. Early changes in plasma amino acid concentrations during aggressive nutritional therapy in extremely low birth weight infants. J Pediatr. 2011 Apr;158(4):543-548.e1. doi: 10.1016/j.jpeds.2010.09.082. Epub 2010 Dec 3. PMID 21129755
- [Derived] Blanco CL, Falck A, Green BK, Cornell JE, Gong AK. Metabolic responses to early and high protein supplementation in a randomized trial evaluating the prevention of hyperkalemia in extremely low birth weight infants. J Pediatr. 2008 Oct;153(4):535-40. doi: 10.1016/j.jpeds.2008.04.059. Epub 2008 Jun 27. PMID 18589451